CLINICAL TRIAL: NCT05533411
Title: A Parallel-group Treatment, Phase 1, Participant- and Investigator-Blind, Randomized Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Intravenous Dose of Donanemab Compared With Placebo in Healthy Chinese Participants
Brief Title: A Study of Donanemab (LY3002813) in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18244; I5T-MC-AACK (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Healthy
MeSH Terms: interventions — donanemab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 350 milligram (mg) Donanemab (Experimental): Single 350 mg Donanemab dose administered intravenously (IV) on Day 1.
  Interventions: Drug: Donanemab
- 700 mg Donanemab (Experimental): Single 700 mg Donanemab dose administered IV on Day 1.
  Interventions: Drug: Donanemab
- 1400 mg Donanemab (Experimental): Single 1400 mg Donanemab dose administered IV on Day 1.
  Interventions: Drug: Donanemab
- Placebo (Placebo Comparator): Single placebo dose administered IV on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donanemab — Administered IV.
  Other Names: LY3002813
  Arms: 1400 mg Donanemab; 350 milligram (mg) Donanemab; 700 mg Donanemab
Drug: Placebo — Administered IV.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of donanemab (LY3002813) when administered as single dose in healthy Chinese participants. The study will also assess how fast donanemab gets into the blood stream and how long it takes the body to remove it. The study is open to healthy participants. The study will last up to approximately 85 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Participants are native Chinese participants. To qualify as a native Chinese, the participant, the participant's biological parents, and all four of the participant's biological grandparents must be of Chinese origin.
* Have a body mass index (BMI) of 18.0 and 28.0, kilograms per meter squared (kg/m²), inclusive.

Exclusion Criteria:

* Are lactating.
* Are women of childbearing potential.
* Have known allergies to donanemab, related compounds or any components of the formulation or history of significant atopy.
* Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within three months or five half-lives (whichever is longer) prior to dosing.
* Have participated, within the last 30 days, in a clinical study involving an investigational product; at least five half-lives or 30 days (whichever is longer) should have passed.
* Have history of intracranial hemorrhage, cerebrovascular aneurysm or arteriovenous malformation, or carotid artery occlusion, stroke or epilepsy.
* Participants who show evidence of positive HIV antibodies, or positive hepatitis C antibody, or positive hepatitis B surface antigen
* Have had leukemia, lymphoma, or any malignancy within the past five years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for three years. Have had breast cancer within the past 10 years.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single placebo dose administered intravenously (IV) on Day 1.
- 350 Milligram (mg) Donanemab: Single 350 mg Donanemab dose administered IV on Day 1.
Period: Overall Study
Arm/Group | Placebo | 350 Milligram (mg) Donanemab | 700 mg Donanemab | 1400 mg Donanemab
Started | 6 | 10 | 10 | 10
Received At Least 1 Dose of Study Drug | 6 | 10 | 10 | 10
Completed | 6 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 350 mg Donanemab: Single 350 mg Donanemab dose administered IV on Day 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | 350 mg Donanemab | 700 mg Donanemab | 1400 mg Donanemab | Total
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (7.0) | 28.1 (6.2) | 32.8 (4.5) | 27.9 (5.8) | 29.2 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 10 | 10 | 10 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 10 | 10 | 10 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 6 | 10 | 10 | 10 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality is located in the Reported Adverse Event module. Drug related TEAEs are any untoward medical occurrences that either occurs postdose or presents prior to dosing yet becomes more severe postdose, and in the opinion of the investigator is possibly related to study drug.
Time Frame: Baseline up to Day 85
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Number; unit: participants
Arm/Group | Placebo | 350 mg Donanemab | 700 mg Donanemab | 1400 mg Donanemab
Number analyzed (Participants) | 6 | 10 | 10 | 10
participants
  Treatment-emergent Adverse Events | 1 | 2 | 0 | 0
  Serious Adverse Events | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Donanemab
Description: PK: Cmax of Donanemab
Time Frame: Predose, Days 2, 3, 4, 5, 8, 15, 22, 29, 43, 57 and 85 postdose
Population: All enrolled participants who received at least 1 full dose of donanemab and had baseline, and at least 1 postbaseline evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | 350 mg Donanemab | 700 mg Donanemab | 1400 mg Donanemab
Number analyzed (Participants) | 10 | 10 | 10
microgram per milliliter (μg/mL) | 119 (13) | 236 (9) | 539 (30)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Donanemab
Description: PK: AUC[0-∞] of Donanemab
Time Frame: Predose, Days 2, 3, 4, 5, 8, 15, 22, 29, 43, 57 and 85 postdose
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: microgram * hour/milliliter (μg.h/mL)
Arm/Group | 350 mg Donanemab | 700 mg Donanemab | 1400 mg Donanemab
Number analyzed (Participants) | 9 | 10 | 10
microgram * hour/milliliter (μg.h/mL) | 9050 (23) | 22600 (17) | 53100 (27)

ADVERSE EVENTS:
Time Frame: Baseline up to 85 days
Description: All participants randomly assigned to study intervention and who take at least 1 dose of study intervention.
Groups:
- 350 Milligrams (mg) Donanemab: Single 350 mg Donanemab dose administered IV on Day 1.
Arm/Group | Placebo | 350 Milligrams (mg) Donanemab | 700 mg Donanemab | 1400 mg Donanemab
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/6 | 6/10 | 4/10 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | 350 Milligrams (mg) Donanemab (N=10) | 700 mg Donanemab (N=10) | 1400 mg Donanemab (N=10)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT05533411/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT05533411/SAP_001.pdf